CLINICAL TRIAL: NCT01427114
Title: Open-labeled, Multicenter Phase II Study of Rituximab, Cyclophosphamide, Vincristine, and Prednisolone (R-CVP) Chemotherapy in Patients With Non-conjunctival Ocular Adnexal MALT Lymphoma
Brief Title: R-CVP for the Treatment of Non-conjunctival Ocular Adnexal MALT Lymphoma (OAML)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Konkuk University Medical Center (Other)
Collaborators: Seoul St. Mary's Hospital (Other)
Responsible Party: Principal Investigator, Sung-Yong Kim, Assistant Professor, Konkuk University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KUH1010258
Record Dates: First submitted 2011-08-30; First posted 2011-09-01 (Estimated); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Lymphoma
Keywords: extranodal marginal zone lymphoma; ocular adnexal lymphoma; mucosa associated lymphoid tissue; cyclophosphamide; vincristine; prednisolone
MeSH Terms: conditions — Lymphoma | interventions — Rituximab; Cyclophosphamide; Vincristine; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- R-CVP (Experimental): 6 cycles of R-CVP followed by 2 cycles of rituximab
  Interventions: Drug: rituximab, cyclophosphamide, vincristine, and prednisolone

INTERVENTIONS:
Drug: rituximab, cyclophosphamide, vincristine, and prednisolone — 6 cycles of R-CVP followed by 2 cycles of rituximab
  Other Names: 6 cycles of R-CVP followed by 2 cycles of rituximab

SUMMARY:
The purpose of this study is to determine how efficient the combination of rituximab, cyclophosphamide, vincristine, and prednisolone (R-CVP) is in the treatment of stage I or II non-conjunctival ocular adnexal MALT lymphoma (OAML).

DETAILED DESCRIPTION:
The treatment of stage I or II OAML is mainly composed of radiotherapy because chemotherapy including cyclophosphamide, vincristine, and prednisolone (CVP) did not show the acceptable response rate compared with radiotherapy. However, radiotherapy for this disease can cause many complications of eyes. This clinical trial was designed to examine the efficacy of R-CVP combination therapy as a first-line treatment for stage I or II non-conjunctival OAML aiming to avoid radiation hazard and increase the efficacy of CVP chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed OAML
* Non-conjunctival or bilateral conjunctival (TNM-based, above T1N0M0 or bT1N0M0), Ann Arbor stage I and II OAML
* Previously untreated
* Age ≥18 years
* Performance status: ECOG 0-2
* Adequate hematological function: hemoglobin ≥9 g/dL,, absolute neutrophil count (ANC) ≥1,500/μL, and platelet count ≥100,000/μL, unless abnormalities are due to bone marrow involvement by the lymphoma
* Adequate liver function tests:

  i. Transaminase (AST/ALT) <3 times the upper normal value ii. Bilirubin <2 times the upper normal value
* Adequate renal function:serum creatinine level <2 mg/dL (177 μmol/L)
* Life expectancy ≥ 6 months
* A negative serum or urine pregnancy test before treatment must be available for both premenopausal women and for women who have <2 years after the onset of menopause.
* Informed consent

Exclusion Criteria:

* NHL subtypes other than OAML
* Primary conjunctival OAML, unilateral involved (T1N0M0)
* Ann Arbor stage III or IV
* CNS involvement by the lymphoma or any evidence of spinal cord compression. Brain CT/MRI is only mandatory (within 4 weeks) with clinical suspicion of CNS involvement by the lymphoma
* Pregnant or lactating women, women of child-bearing potential not using adequate contraception
* Inadequate liver function tests:

  i. Transaminase (AST/ALT) ≥3 times the upper normal value or ii. Bilirubin ≥2 times the upper normal value
* Inadequate renal function:

  i. serum creatinine level <2 mg/dL (177 μmol/L)
* Other serious illness or medical conditions i. Unstable cardiac disease despite treatment; myocardial infarction within 6 months prior to study entry ii. History of significant neurological or psychiatric disorders including dementia or seizures
* Active uncontrolled infection (HIV, hepatitis B, Hepatitis C, active Tuberculosis, active bacterial, or active fungal infection)
* Any other malignancies within the past 5 years except for curatively treated non-melanoma skin cancer or in situ carcinoma of the cervix uteri
* Known hypersensitivity to any of the study drugs or its ingredients (i.e., hypersensitivity to Polysorbate 20, CHO cell products, or recombinant human antibodies)
* Concomitant administration of any other experimental drug under investigation or concomitant chemotherapy, hormonal therapy, or immunotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-07-01 (Actual); Primary Completion 2014-08-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
complete response rate | 3 years
  CR rate

SECONDARY OUTCOMES:
Progression free survival | 5 years
  Progression free survival
Overall survival | 5 years
  Overall survival
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 5 years
  Number of Participants with Adverse Events as a Measure of Safety and Tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Seok-Goo Cho, Ph.D., Principal Investigator — Seoul St. Mary's Hospital; Sung-Yong Kim, Ph.D., Principal Investigator — Konkuk University Medical Center
Locations (2):
- South Korea (2):
  - Seoul St. Mary's Hospital, Seoul
  - KonKuk University Medical Center, Seoul

REFERENCES:
- [Derived] Kim SY, Yang SW, Lee WS, Yang JW, Oh SY, Ahn HB, Yang DH, Park SK, Chang JH, Kim HJ, Lee MJ, Cho SG. Frontline treatment with chemoimmunotherapy for limited-stage ocular adnexal MALT lymphoma with adverse factors: a phase II study. Oncotarget. 2017 Aug 2;8(40):68583-68590. doi: 10.18632/oncotarget.19788. eCollection 2017 Sep 15. PMID 28978139